CLINICAL TRIAL: NCT01520025
Title: Direct Imaging of Ischemia With 18F-FDG PET Imaging Combined With Coronary Anatomy From CT Coronary Angiography
Brief Title: Multi-modality Imaging of Ischemia With 18F-FDG PET and CTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Continued recruitment of study participants was not feasible
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Principal Investigator, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HI Protocol #2011397-01H
Record Dates: First submitted 2011-07-15; First posted 2012-01-27 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Myocardial Ischemia
Keywords: Radiopharmaceutical; 18FDG PET; CTA; Multi-modality imaging; Metabolic Imaging of Ischemia; Myocardial blood flow; Myocardial blood flow reserve
MeSH Terms: conditions — Myocardial Ischemia | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG PET imaging (Experimental): Positron Emission Tomography nuclear stress scan following either pharmacologic or treadmill stress test with radiopharmaceutical injection at peak stress or within 1 hour following peak stress.
  Interventions: Radiation: PET MPI imaging with 18F-Fluorodeoxyglucose

INTERVENTIONS:
Radiation: PET MPI imaging with 18F-Fluorodeoxyglucose — Exercise Stress Testing. All patients will undergo a symptom-limited exercise treadmill test using the Bruce protocol after a 24 hour high fat, low carbohydrate diet and an overnight fast. Persantine Stress Testing: Subjects who have undergone Persantine stress protocol for the PET or SPECT will follow the same protocol. A high fat, low carbohydrate diet for 24 hours and a 12 hour overnight fast will precede the study stress scan. Anti-anginal medications will be withheld on the morning of the exercise test.
  18FDG (370 mBq) will be injected at either peak exercise or within 1 hour of peak.
  Patients will be imaged 60 minutes after radiotracer injection in the supine position in a Discovery 690/VCTLYSO PET system (GE Healthcare, Milwaukee, Wisconsin)

SUMMARY:
Coronary artery disease results in narrowing of the blood vessels supplying oxygenated blood to the heart muscle. Diagnosis in patients with symptoms of chest pain is now quickly done with CT coronary angiography. This x-ray test can show narrowed blood vessels but has limited ability to predict the severity of the narrowings in some cases. We have described a new approach using PET exercise 18F-FDG imaging as a method to image areas of heart muscle not getting enough blood during exercise stress. The 18F-FDG images are co-registered with the CT anatomy from the CTA to provide direct evidence of the consequences of the narrowing.

DETAILED DESCRIPTION:
The Investigators and others have demonstrated direct imaging of myocardial ischemia using 18F-Fluorodeoxyglucose (18FDG) with exercise or dipyridamole stress and positron emission tomography (PET) or single photon emission computed tomography (SPECT). This approach with "hot-spot" imaging may have greater diagnostic accuracy for ischemia than conventional "cold-spot" myocardial perfusion imaging.

Recent advances in multi-modality imaging permit fusion of CTA images with PET or SPECT perfusion images and functional assessment of anatomical CAD. Registration of the 2 data sets can be optimized using the CT acquired with the PET or SPECT15. 18FDG uptake as a marker for ischemia can be directly related to the coronary anatomy and guide revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected CAD referred for CTA and found to have moderate CAD stenoses and 20 normal volunteers with less than 5% probability of CAD.
2. Age ≥ 18 years

Exclusion Criteria:

1. Inability to undergo stress protocol due to co-morbidities
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Extent of ischemia as determined by visual and quantitative analysis | at time of scan

SECONDARY OUTCOMES:
The degree of correlation between the multiple modalities (CTAm stress PET or SPECT and 18FDG PET) | 3 to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Abramson BL, Ruddy TD, deKemp RA, Laramee LA, Marquis JF, Beanlands RS. Stress perfusion/metabolism imaging: a pilot study for a potential new approach to the diagnosis of coronary disease in women. J Nucl Cardiol. 2000 May-Jun;7(3):205-12. doi: 10.1016/s1071-3581(00)70008-0. PMID 10888390
- [Background] He ZX, Shi RF, Wu YJ, Tian YQ, Liu XJ, Wang SW, Shen R, Qin XW, Gao RL, Narula J, Jain D. Direct imaging of exercise-induced myocardial ischemia with fluorine-18-labeled deoxyglucose and Tc-99m-sestamibi in coronary artery disease. Circulation. 2003 Sep 9;108(10):1208-13. doi: 10.1161/01.CIR.0000088784.25089.D9. Epub 2003 Aug 25. PMID 12939208
- [Background] Abbott BG, Liu YH, Arrighi JA. [18F]Fluorodeoxyglucose as a memory marker of transient myocardial ischaemia. Nucl Med Commun. 2007 Feb;28(2):89-94. doi: 10.1097/MNM.0b013e328013eaa5. PMID 17198348